CLINICAL TRIAL: NCT06063733
Title: Development and Feasibility Testing of Digital Theory-based Pursed Lip Breathing in Stable Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Houqiang Huang, A postgraduate researcher in the School of Nursing & Public Health, Manchester Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KY2023105
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pursed lip breathing; Behavioral interventions; Gamification
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital PLB intervention (Experimental): Participants will perform the following tasks during the intervention:
  1. Register a personal account on the theory-based pursed lip breathing intervention protocol software system installed on smartphones(DT-PLB).
  2. Acquire knowledge and skills related to pursed lip breathing by watching instructional videos.
  3. Practice Pursed Lip Breathing for 10 minutes per session, three times daily for eight weeks, as per reminders and guidance provided by the software.
  4. Earn health points by completing specific actions as instructed.
  5. Optionally post individual texts on the peer forum for peer support within the DT-PLB software.
  6. Complete two outcome assessments as scheduled.
  Interventions: Other: Digital pursed lip breathing intervention

INTERVENTIONS:
Other: Digital pursed lip breathing intervention — After registration, participants will watch an educational video on the developed software, covering the definition, benefits, and techniques of pursed lip breathing. Following this, participants will engage in pursed lip breathing interventions, guided by voice and animated instructions from the software. These sessions will occur three times daily (morning, afternoon, and night) for 10 minutes each, lasting for 8 weeks.
  After each session, participants can choose to post texts on a peer social forum for peer support. Fellow participants can give 'comments' or 'likes'. The principal researcher will oversee texts, peer comments, removing information containing personal data, medical recommendations, and negative comments.
  Additionally, participants can earn health points by performing specific actions (e.g., watching the educational video and practicing pursed lip breathing) on the software, encouraging their participation in related activities.

SUMMARY:
The goal of this pre-post design clinical trial is to develop a digital, theory-based Pursed Lip Breathing intervention protocol software system installed on smartphones (DT-PLB) and to preliminarily evaluate its feasibility and effects in stable Chronic Obstructive Pulmonary Disease (COPD). The main objectives are:

1. To develop a digital, theory-based Pursed Lip Breathing intervention protocol software system installed on smartphones for managing breathing exercises in stable COPD patients.
2. To pilot the methodological procedures of the pre-post study.
3. To determine the recruitment rate, retention rate, attrition rate, and software usage compliance during the subject recruitment and follow-up process of the pre-post study.
4. To evaluate the perception and satisfaction of COPD patients using the DT-PLB.
5. To preliminarily examine the effects of using the DT-PLB intervention on COPD patients, including the six-minute walking test, FEV1% predicted, FEV1/FVC, mMRC scale, COPD assessment test scale, and health points.
6. To identify any potential adverse events associated with the implementation of DT-PLB.

Participants will perform the following tasks during the intervention:

1. Register a personal account on the DT-PLB software.
2. Acquire knowledge and skills related to Pursed Lip Breathing by watching instructional videos.
3. Practice Pursed Lip Breathing for 10 minutes per session, three times daily for eight weeks, as per reminders and guidance provided by the software.
4. Earn health points by completing specific actions as instructed.
5. Optionally post individual texts on the peer forum for peer support within the DT-PLB software.
6. Complete two outcome assessments as scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD satisfying GOLD criteria (Agusti, 2022) ;
* Being Chinese;
* Able to understand, speak, and hear;
* Clinically stable for at least three months prior to enrollment (Soler-Cataluna et al., 2018) ;
* The classification of GOLD grades for patients is mild, moderate, and severe, which means: FEV1/FVC<70%, FEV1>30%pre (Agusti, 2022) ;
* Participants who were mindful about the IT technology and known how to use a smartphone.

Exclusion Criteria:

* Impaired hand function causing inability to use the application;
* Have disorders in pleural effusion, pulmonary malignancy, heart diseases, stroke with sequels;
* Patients who have oral or nasal diseases cannot complete the exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of participants who participate in the study divided by the number of participants eligible for participation
Retention rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of subjects who complete the study divided by the number of subjects who participate in the study
Attrition rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of subjects who drop out after participation divided by the number of subjects who participate in the study
Software usage Compliance | Immediately after completion of the 8-week intervention
  The compliance rate is one of compliance outcomes, reflecting the level of patient engagement in the intervention. Overall compliance will be defined as the compliance averaged in all patients. Compliance rate = (actual number of participation in the intervention/planned number of sessions)x 100%. In addition, minutes-consuming recorded on the software for participants during the research will be used to complement outcome measures of compliance.
Adverse events associated with the DT-PLB intervention | Immediately after completion of the 8-week intervention
  In each DT-PLB session, the participants during the intervention will record whether they had any uncomfortable feelings

SECONDARY OUTCOMES:
mMRC Dyspnea Scale | From baseline (T1) to the completion of the 8-week intervention (T2)
  The Modified Medical Research Council (mMRC) Dyspnea Scale consists of five categories, ranging from 0 to 4, with higher scores indicating more severe breathlessness. A score of 0 indicates no breathlessness during activities, while a score of 4 suggests breathlessness.
CAT scale | From baseline (T1) to the completion of the 8-week intervention (T2)
  COPD assessment test (CAT)is a questionnaire-based tool that is commonly used to assess the impact of chronic obstructive pulmonary disease (COPD)on a patient's health status and quality of life. It consists of eight questions that cover a range of symptoms, including cough, sputum production, breathlessness, chest tightness, and activity limitations. Each question on the CAT is scored on a scale from 0 to 5, with a maximum possible score of 40. A higher score indicates a greater degree of symptom severity and a poorer health status.
The System Usability Scale | Immediately after completion of the 8-week intervention (T2)
  The system usability scale (SUS)is a standardized questionnaire that is used to evaluate the usability and user experience of a wide range of products, services, and systems. It produces a score between 0 and 100, with higher scores indicating better usability and user experience. The SUS has been validated and is widely used in both industry and research settings to evaluate the usability and user experience of a wide range of systems and products, including software applications, websites, and medical devices.
Participants overall satisfaction | Immediately after completion of the 8-week intervention (T2)
  Participants will be required to rate their satisfaction with this software intervention, with a 10-point numeric rating scale (NRS) , where "1" represents "very dissatisfied" and "10" means "very satisfied".
Six-minute-walking test | From baseline (T1) to the completion of the 8-week intervention (T2)
  The Six-Minute Walk Test is a commonly used measure of functional exercise
Pulmonary function index:FEV1%predicted, FEV1/FVC | From baseline (T1) to the completion of the 8-week intervention (T2)
  FEV1%predicted stands for "forced expiratory volume in one second predicted" and is a measure of lung function. It represents the maximum amount of air that a person can forcefully exhale from their lungs in one second. FEV1%predicted is expressed as a percentage of the predicted value for someone with the same characteristics who does not have lung disease.
  FEV1/FVC is another measure of lung function, which represents the ratio of the amount of air that a person can forcefully exhale in one second (FEV1)to the total amount of air that they can exhale(forced vital capacity or FVC)over the course of a full exhalation. A low FEV1/FVC ratio indicates that the airways are obstructed or narrowed, which is a characteristic feature of COPD.
Health points obtained by each participant performing formulated operations | Immediately after completion of the 8-week intervention
  Health points are set based on consensus, obtained by operating actions on this software:
  1. Login: participants' stay on the software lasts for over one minute, they will earn one health point, with a maximum of three health points per day.
  2. Watch PLB health education video: For every minute participants stay on the video, they will earn one health point. The maximum score for a single viewing is equal to the length of the video.
  3. Accept PLB exercise task: Earning one health point upon claiming an exercise task. For every minute spent on the exercise animated videos, patients earn one health point, with a maximum of up to ten health points.
  4. Social forum: Participants can post an update in an internal forum, earning them one health point, with a maximum of three health points per day.
  5. Reward health points of consecutive accepted tasks: an additional rewarded 50 points for continuously claiming exercises tasks for 9 consecutive times.

CONTACTS AND LOCATIONS:
Overall Officials: Houqiang Huang, Master, Principal Investigator — Manchster Metropolitan University
Locations (1):
- The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang H, Liu F, Mohammad M, Watson R, Hayter M, Huang M, Li Z. Digital gamification-based pursed lip breathing exercises driven by Behaviour Change Wheel in patients with COPD: a feasibility trial protocol using pre-post study design. BMJ Open. 2025 Mar 27;15(3):e090832. doi: 10.1136/bmjopen-2024-090832. PMID 40147988